CLINICAL TRIAL: NCT05720364
Title: A Phase 1, Open-Label, Randomized, Single-Dose, Parallel-Group Study to Evaluate the Food Effect on the Pharmacokinetics of TP-05 Under Fed and Fasted Conditions in Healthy Participants
Brief Title: Study to Evaluate the Food Effect of TP-05 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRS-017
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — lotilaner

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TP-05, Fasted Group (Experimental): Single dose of TP-05 (lotilaner oral), fasted
  Interventions: Drug: TP-05 (lotilaner oral), fasted group
- TP-05, High-Fat Group (Experimental): Single dose of TP-05 (lotilaner oral) following a high-fat meal
  Interventions: Drug: TP-05 (lotilaner oral), high-fat group
- TP-05, Low-Fat Group (Experimental): Single dose of TP-05 (lotilaner oral) following a low-fat meal
  Interventions: Drug: TP-05 (lotilaner oral), low-fat group

INTERVENTIONS:
Drug: TP-05 (lotilaner oral), fasted group — TP-05 (lotilaner oral), fasted group
  Other Names: TP-05, fasted
  Arms: TP-05, Fasted Group
Drug: TP-05 (lotilaner oral), high-fat group — TP-05 (lotilaner oral), high-fat group
  Other Names: TP-05, high-fat meal
  Arms: TP-05, High-Fat Group
Drug: TP-05 (lotilaner oral), low-fat group — TP-05 (lotilaner oral), low-fat group
  Other Names: TP-05, low-fat meal
  Arms: TP-05, Low-Fat Group

SUMMARY:
A Phase 1, Open-Label, Randomized, Single-Dose, Parallel-Group Study to Evaluate the Food Effect on the Pharmacokinetics of TP-05 under Fed and Fasted Conditions in Healthy Participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, single-dose, parallel-group study to evaluate the food effect on the pharmacokinetics of TP-05 under fed and fasted conditions in healthy participants.

The study will consist of a screening period of up to 28 days. Participants who are eligible for the study will check into the clinical research site on Day -1. All participants will undergo an overnight fast of at least 10.5 hours prior to dosing. On Day -1 participants will be randomized to receive one of three treatment regimens on Day 1: single dose of TP-05, fasted; single dose of TP-05 following a high-fat breakfast; or single dose of TP-05 following a low-fat breakfast.

Participants will be resident at the clinical research site from Day -1 until completion of assessments at 96 hours post-dose (Day 5) and return on Day 60 for a follow-up visit. Participants will complete a telephone safety follow-up visit at Day 120.

Safety will be assessed by adverse events, vital signs, performing physical examinations, electrocardiograms, and evaluating clinical laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history and physical examination
* Participants who are non- or ex-smokers
* No clinically significant disease captuired in medical history or evidence of clinically significant findings on the physical examination and/or ECG at Screening and Day -1, as determined by the Investigator
* BMI 18.5-29.9 kg/m2 (inclusive) and weighs at least 50.0 kg at Screening
* Ability to comply with contraceptive requirements

Exclusion Criteria:

* Female who is breast-feeding or pregnancy according to the serum pregnancy test at Screening and urine pregnancy test at Day -1 prior to study drug administration
* History of significant hypersensitivity to lotilaner or any related products
* History of significant gastrointestinal, metabolic, liver, or kidney disease, or surgery that may affect drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
* History of malignancy (or active malignancy), with the exception of treated basal cell or squamous cell carcinoma
* Positive test results for HIV-1/HIV-2 antigen/antibody, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb)
* Positive result for SARS-CoV-2 testing at Day -1
* Use of any non-prescription or prescription drugs in the 7 days or 5 half-lives (whichever is longer) prior to study drug administration and through the treatment period of the study
* Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to Screening and through Day 60 of the study
* History of live attenuated vaccine within 4 weeks prior to study drug administration or requirement to receive these vaccinations through Day 60 of the study
* Plasma donation within 7 days prior to Screening through Day 60 of the study
* Blood donation or significant blood loss approximately 500 mL within 56 days prior to Screening through Day 60 of the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Concentration of TP-05 in whole blood | Up to Day 60
  PK parameters for whole blood sampling methods following dose administration with a high-fat meal, low-fat meal, and fasting will be evaluated. Parameter includes concentration level.
Exposure and PK of lotilaner in whole blood (AUC0-96hours) | Up to Day 5
  PK parameters for whole blood sampling methods following dose administration with a high-fat meal, low-fat meal, and fasting will be evaluated. Parameter includes AUC0-96hours.
Exposure and PK of lotilaner in whole blood (Cmax) | Up to Day 60
  PK parameters for whole blood sampling methods following dose administration with a high-fat meal, low-fat meal, and fasting will be evaluated. Parameter includes Cmax.
Exposure and PK of lotilaner in whole blood (Tmax) | Up to Day 60
  PK parameters for whole blood sampling methods following dose administration with a high-fat meal, low-fat meal, and fasting will be evaluated. Parameter includes Tmax.
Exposure and PK of lotilaner in whole blood (Tlag) | Up to Day 60
  PK parameters for whole blood sampling methods following dose administration with a high-fat meal, low-fat meal, and fasting will be evaluated. Parameter includes Tlag.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to Day 120
  Evaluate the safety of TP-05 through the incidence rate of TEAEs
Clinically significant changes from Baseline chemistry laboratory tests | Up to Day 60
  Evaluate the safety of TP-05 through clinically significant changes from Baseline chemistry laboratory tests
Clinically significant changes from Baseline physical examination | Up to Day 60
  Evaluate the safety of TP-05 through clinically significant changes from Baseline physical examinations
Clinically significant changes from Baseline vital signs | Up to Day 60
  Evaluate the safety of TP-05 through clinically significant changes from Baseline vital signs
Clinically significant changes from Baseline electrocardiograms (ECGs) | Up to Day 60
  Evaluate the safety of TP-05 through clinically significant changes from Baseline ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Jose Trevejo, MD, PhD, Study Director — Tarsus Pharmaceuticals, Inc.
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States